CLINICAL TRIAL: NCT04511910
Title: How to Predict Postoperative Complications After Early Laparoscopic Cholecystectomy for Acute Cholecystitis: the Chole-Risk Score
Acronym: CholeRiskScore
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Marcello Di Martino (Unknown)
Responsible Party: Sponsor
Other Study IDs: CholeRisk Score
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2020-12

CONDITIONS: Cholecystitis, Acute
Keywords: Acute cholecystitis; Cholecystectomy; Gallbladder
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early surgery Group 1: The surgery is performed within the first 3 days
  Interventions: Procedure: Early Laparoscopic Cholecystectomy
- Early surgery Group 2: Surgery is performed between the fourth and seventh day
  Interventions: Procedure: Early Laparoscopic Cholecystectomy
- Early surgery Group 3: Surgery is performed more than 7 days from the onset of symptoms
  Interventions: Procedure: Early Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Early Laparoscopic Cholecystectomy

SUMMARY:
Acute calculous cholecystitis (ACC) is the most common complication of gallstone disease, and laparoscopic cholecystectomy is the gold standard treatment. Several prospective studies have demonstrated that same-admission, early LC (ELC), for ACC is safe when compared with delayed LC (DLC). However, there is still controversy on the indication of ELC in high risk patients with important comorbidities, in cases of severe inflammation of the gallbladder and in patients with ACC and suspicious of a choledocholithiasis. The advantages of ELC in high risk patients with severe comorbidities have been recently questioned, with Tokyo Guidelines 2018 (TG18) proposing an initial conservative management of this cases, assessing the benefit of ELC according to specified criteria. However, the recent CHOCOLATE trial, demonstrated the advantages of ELC over an initial conservative management. Performing an ELC for ACC can be a straightforward procedure for an on-call general surgeon or a very challenging procedure even for experienced hepatopancreaticobiliary (HPB) laparoscopic surgeon, depending on disease features, surgeons experience, centres volumes and resources available. Deciding whether the ELC should be performed by the on-call team or by HPB surgical team, or whether the operation should be delayed are still matter of debate in daily practice.

Several preoperative scores assessing the risk of difficult cholecystectomy have been proposed, but they were mainly focused on elective procedures and on risk of conversion to open cholecystectomy or other intraoperative complications. They did not asses the risk of post-operative complications in a subgroup of patients, for whom, indication to ELC by the on-call general surgeon is still questionable according to the more recent guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed with Acute calculous cholecystitis.
* Consecutive patients undergoing early laparoscopic cholecystectomy between January 2013 and December 2018 during admission for the acute episode.
* Minimum 30-day post-operative follow-up.
* ASA ≤ 3.

Exclusion Criteria:

* Presence of another concomitant pathology of the bile duct (choledocholithiasis, cholangitis, pancreatitis, biliary peritonitis).
* Aetiology other than cholelithiasis (amythiasis, malignancy).
* Patients with severe sepsis, immunosuppression and pregnancy.
* Additional abdominal surgical procedure.
* ASA 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLP surgery patients between January 2013 and December 2018. The diagnosis of acute cholecystitis will be established according to the Tokio Guidelines:
  * Local signs (pain in right hypochondrium / Murphy's sign).
  * Systemic (fever / elevated C-reactive protein / leukocytosis)
  * Ultrasound findings (gallbladder distension, wall thickening, pericolectic fluid or radiological Murphy's sign, associated with gallstones). In all patients, treatment with antibiotics will be carried out according to each hospital's protocols in terms of type and duration.
Sampling Method: Non-Probability Sample
Enrollment: 1868 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Increased post-operative complications | For at least 30 postoperative days
  Patients who only developed Clavien-Dindo I-II complications were assigned to group 1 (G1), whereas groups 2 (G2) included patients with post-operative complications ≥ IIIa. Patients with post-operative LOS greater than 10 days and who required readmissions within 30 days from the discharge were also assigned to G2.
Number of Participants with Postoperative hemorrhagia | For at least 30 postoperative days
  Postoperative hemorrhagia
Number of Participants with Biliary fistula | For at least 30 postoperative days
  Biliary fistula
Number of Participants with Jaundice | For at least 30 postoperative days
  Jaundice
Number of Participants with Cardiac insufficiency | For at least 30 postoperative days
  Cardiac insufficiency
Number of Participants with Heart infarction | For at least 30 postoperative days
  Heart infarction
Number of Participants with Respiratory insufficiency | For at least 30 postoperative days
  Respiratory insufficiency
Number of Participants with Pulmonary thromboembolism | For at least 30 postoperative days
  Pulmonary thromboembolism
Number of Participants with Kidney failure or dialysis | For at least 30 postoperative days
  Kidney failure or dialysis

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital Universitario German Trias I Pujol, Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Cruces, Bilbao, Vizcaya
  - Hospital Universitario de la Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No